CLINICAL TRIAL: NCT06072781
Title: A Phase 3, Randomized, Open-Label Study of Combination Therapy With Avutometinib Plus Defactinib Versus Investigator's Choice of Treatment in Patients With Recurrent Low-Grade Serous Ovarian Cancer (LGSOC) (RAMP 301)
Brief Title: A Study of Avutometinib (VS-6766) + Defactinib (VS-6063) in Recurrent Low-Grade Serous Ovarian Cancer
Acronym: RAMP 301
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Australia New Zealand Gynaecological Oncology Group (Other); Korean Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-301; GOG-3097 (Other: The GOG Foundation, Inc.); ENGOT-ov81 (Other: ENGOT)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Low Grade Serous Ovarian Cancer
Keywords: Low Grade Serous Ovarian Cancer; KRAS; KRAS wt; KRAS mt
MeSH Terms: interventions — defactinib; liposomal doxorubicin; Paclitaxel; Letrozole; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- avutometinib + defactinib (Experimental): Avutometinib 3.2 mg, PO, twice weekly for 21 days on, 7 days off in a 28-day (4 weeks) cycle in combination with defactinib 200 mg, PO, twice daily for 21 days on, 7 days off in a 28-day(4 week) cycle.
  Interventions: Drug: avutometinib; Drug: Defactinib
- Investigator Choice of Treatment (ICT) (Active Comparator): Patients will receive one of the following therapies as determined by the Investigator:
  * Pegylated liposomal doxorubicin: 40 mg/m2 IV on Day 1 of each 28-day (4 week) cycle.
  * Paclitaxel: 80 mg/m2 IV on Days 1, 8, and 15 of each 28-day (4 week) cycle.
  * Anastrozole: 1 mg, PO, once daily of each 28-day (4 week) cycle.
  * Letrozole: 2.5 mg, PO, once daily of each 28-day (4 week) cycle.
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Paclitaxel; Drug: Letrozole; Drug: Anastrozole

INTERVENTIONS:
Drug: avutometinib — Avutometinib: administered orally
  Other Names: avutometinib (VS-6766)
  Arms: avutometinib + defactinib
Drug: Defactinib — Defactinib: administered orally
  Other Names: defactinib (VS-6063)
  Arms: avutometinib + defactinib
Drug: Pegylated liposomal doxorubicin — administered intravenously
  Other Names: Caelyx, Doxil, Lipodox
  Arms: Investigator Choice of Treatment (ICT)
Drug: Paclitaxel — administered intravenously
  Other Names: Nov-Onxol, Onxol, Navaplus, Taxol
  Arms: Investigator Choice of Treatment (ICT)
Drug: Letrozole — administered orally
  Other Names: Femara
  Arms: Investigator Choice of Treatment (ICT)
Drug: Anastrozole — administered orally
  Other Names: Arimidex
  Arms: Investigator Choice of Treatment (ICT)

SUMMARY:
This study will assess the safety and efficacy of avutometinib (VS-6766) in combination with defactinib versus Investigator's choice of treatments (ICT) in subjects with recurrent LGSOC who have progressed on a prior platinum-based therapy.

DETAILED DESCRIPTION:
This international, randomized, open-label, Phase 3 study will compare the investigational combination of avutometinib plus defactinib versus Investigator's Choice of Treatments (ICT) in patients with recurrent LGSOC who have progressed on a prior platinum-based therapy. Avutometinib and defactinib are both types of drugs called kinase inhibitors. Kinase inhibitors block cancer cell growth. The study will compare the progression-free survival (PFS) of the combination of avutometinib plus defactinib versus ICT. The study will also evaluate the effect of the combination on safety, overall survival, other efficacy endpoints, and health-related quality of life and disease related symptoms. The study is being conducted by gynecological cancer specialists. Patients who are eligible and agree to participate in this study will be treated with either a combination of avutometinib with defactinib, or with one of four standard of care NCCN and ESMO treatment recommendations for recurrent LGSOC, and then with subsequent follow up appointments. Patients who originally received one of the standards of care treatments who are determined to have progressive disease may be eligible to crossover to receive the investigational combination avutometinib plus defactinib.Avutometinib and defactinib are investigational drugs that have not been approved by the U.S. Food and Drug Administration (FDA)

ELIGIBILITY:
Inclusion Criteria:

Patients may be eligible for inclusion in the study if they meet the following criteria:

1. Histologically proven LGSOC (ovarian, fallopian, peritoneal)
2. Documented mutational status of KRAS by a validated tumor-tissue based diagnostic test.
3. Suitable for treatment with at least one of the Investigator's Choice of Treatments:pegylated liposomal doxorubicin, paclitaxel, letrozole, anastrozole.
4. Progression or recurrence of LGSOC after at least one prior systemic therapy for metastatic disease.
5. Measurable disease according to RECIST v1.1.
6. An Eastern Cooperative Group (ECOG) performance status ≤ 1.
7. Adequate organ function.
8. Adequate recovery from toxicities related to prior treatments.
9. For patients with reproductive potential, a negative pregnancy test must be confirmed and agreement to use highly effective method of contraceptive.
10. Willingness to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Systemic anti-cancer therapy within 4 weeks of the first dose of study therapy.
2. Co-existing high-grade serous ovarian cancer or mixed histology.
3. Prior treatment with avutometinib, defactinib, or other FAK inhibitors.
4. History of prior malignancy with recurrence <3 years from the time of enrollment.
5. Major surgery within 4 weeks, minor surgery within 1 week, or palliative radiotherapy within 1 week of the first dose of study intervention.
6. Symptomatic brain metastases requiring steroids or other interventions, known leptomeningeal metastases, or spinal cord compression.
7. An active skin disorder that has required systemic therapy within one year of the first dose of study intervention.
8. History of medically significant rhabdomyolysis.
9. For subjects with prior MEK or RAF exposure, Grade 4 toxicity is deemed related to the MEK inhibitor.
10. Symptomatic bowel obstruction within 3 months of the first dose of study intervention
11. Concurrent ocular disorders.
12. Concurrent heart disease or severe obstructive pulmonary disease.
13. Active or past medical history of interstitial lung disease/pneumonitis, including drug-induced or radiation pneumonitis, pulmonary fibrosis, or adult respiratory distress syndrome (ARDS).
14. Subjects with the inability to swallow oral medications.
15. History of hypersensitivity to any of the active agents or ingredients of study intervention: peanut, soya, polyoxyl castor oil, etcetc.). Prior hypersensitivity to anthracyclines or anthracenediones if the use of pegylated liposomal doxorubicin (PLD) is planned.
16. Pregnant or breastfeeding.
17. Active, uncontrolled infection (bacterial, viral, or fungal) requiring systemic therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2031-02-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per blinded independent central review (BICR) | Up to 24 months
  Progression-free survival (PFS) according to RECIST version 1.1, per blinded independent central review (BICR)

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  From the time of first dose of study intervention to PD as assessed per RECIST 1.1 or death from any cause
Progression Free Survival (PFS) per investigator assessment | 24 months
  Progression-free survival (PFS) according to RECIST version 1.1, per blinded independent central review (BICR)
Objective response rate (ORR) | 12 months
  From the time of first dose of study intervention to PD as assessed per RECIST 1.1 by Investigator or death from any cause
Duration of Response (DOR) | 12 months
  From the time of first dose of study intervention to PD as assessed per RECIST 1.1 by Investigator or death from any cause
Disease Control Rate (DCR) | 6 months
  CR+PR+Stable disease
Frequency and severity adverse events (AEs) and Serious Adverse Events (SAEs) | 25 months
  Count of AE and SAEs by grade, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale
Area under the plasma concentration-time curve (AUC) of avutometinib, defactinib and relative metabolites | 5 months
  Area under plasma Concentration (AUC) 0 to t
Maximum plasma concentration (Cmax) of avutometinib, defactinib and relative metabolites | 5 months
  maximum plasma concentration
To assess the health-related quality of life and disease based on European Organization for Research and Treatment of Cancer (EORTC) Quality of life Questionnaire Core module C30 (QLQ-C30). | 24 months
  The EORTC QLQ-C30 is a validated questionnaire to assess the quality of life of ovarian cancer patients.
To assess the health-related quality of life and disease based on European Organization for Research and Treatment of Cancer (EORTC) Quality of life Questionnaire Ovarian Cancer module OV28 (QLQ-OV28). | 24 months
  The EORTC QLQ-OV28 is a validated questionnaire to assess the quality of life of ovarian cancer patients.
To assess the health-related quality of life and disease based on EuroQol-5 Dimension 5-level (EQ-5D-5L) | 24 months
  The EuroQol-5 Dimension 5-level (EQ-5D-5L) is a validated questionnaire used to measure a patient's overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grisham, MD, Principal Investigator — GOG Foundation; Susana Banerjee, MBBS, MA, PhD, Principal Investigator — European Network of Gynecological Oncological Trial Groups (ENGOT); Craig Berman Verastem Medical Monitor, Study Director — RAMP301@verastem.com
Locations (106):
- United States (38):
  - HonorHealth, Phoenix, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - UCLA Health, Los Angeles, California
  - UC Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Mount Sinai, Miami Beach, Florida
  - AdventHealth, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists Research East, West Palm Beach, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Karmanos Cancer Center, Detroit, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State, Hilliard, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Asplundh Cancer Pavilion | Jefferson Health, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Texas Oncology Central, Austin, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - Houston Methodist, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, San Antonio, Texas
  - Texas Oncology, The Woodlands, Texas
  - Texas Oncology, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
- Australia (5):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (2):
  - UZA, Edegem
  - University Hospital Ghent, Ghent
- Canada (4):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - British of Columbia, Vancouver
- Aalborg U.H, Aalborg, Denmark
- France (5):
  - Centre Hospitalier de Besançon, Besançon
  - Site Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
- Germany (7):
  - Agaplesion Markus Krankenhaus, Frankfurt am Main, Hesse
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Kliniken Essen-Mitte, Essen
  - UMC Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Universitätsfrauenkinik Ulm, Ulm
- St. James's Hospital, Dublin, Ireland
- Italy (12):
  - Centro di Riferimento Oncologico (CRO), Aviano
  - Spedali Civili, Brescia
  - AO Cannizzaro, Catania
  - San Raffaele Hospital, Milan
  - Humanitas San Pio X, Milan
  - European Institute of Oncology (IEO), Milan
  - Istituto Nazionale dei Tumori, Milan
  - INT Napoli Hospital, Napoli
  - Istituto Oncologico Veneto (IOV), Padua
  - IRCCS Gemelli, Roma
  - Istituti Fisioterapici Ospitalieri, Rome
  - S.C.D.U. Oncologia, Torino
- Japan (5):
  - The Mie University Hospital, Tsu, Mie-ken
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Tohoku University Hospital, Miyagi
  - Osaka Medical Center, Osaka
  - The Jikei University Hospital, Tokyo
- Netherlands (2):
  - Netherlands Cancer Insitute, Amsterdam
  - Radboud UMC, Nijmegen
- Auckland City Hospital, Auckland, New Zealand
- Poland (3):
  - Białostockie Centrum Onkologii, Bialystok
  - Gdański Uniwersytet Medyczny, Gdansk
  - Siedleckie Centrum Onkologii, Siedlce
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam
  - Yonsei University Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Clínico Virgen de La Arrixaca, El Palmar, Murcia
  - H. de Donostia, Donostia / San Sebastian, San Sebastian
  - H. Vall d´ Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - H.U. Ramón y Cajal, Madrid
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (8):
  - Greater Glasgow and Clyde (GGC), Glasgow, Scotland
  - Cambridge University Hospital, Cambridge
  - University of Edinburgh Cancer Research Centre, Edinburgh
  - Hope Cancer Trials Centre, Leicester
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Banerjee SN, Van Nieuwenhuysen E, Aghajanian C, D'Hondt V, Monk BJ, Clamp A, Prendergast E, Oaknin A, Ring K, Colombo N, Holloway RW, Rodrigues M, Chon HS, Gourley C, Santin AD, Thaker PH, Gennigens C, Newman G, Salinas E, Youssoufian H, Moore KN, Lustgarten S, O'Malley DM, Van Gorp T, Grisham RN. The combination of avutometinib and defactinib in treating recurrent low-grade serous ovarian cancer: a plain language summary of the Phase II clinical trial ENGOT-OV60/GOG-3052/RAMP 201. Future Oncol. 2025 Dec;21(30):3859-3871. doi: 10.1080/14796694.2025.2595130. Epub 2025 Dec 12. PMID 41384753
- [Derived] Banerjee SN, Van Nieuwenhuysen E, Aghajanian C, D'Hondt V, Monk BJ, Clamp A, Prendergast E, Oaknin A, Ring K, Colombo N, Holloway RW, Rodrigues M, Chon HS, Gourley C, Santin AD, Thaker PH, Gennigens C, Newman G, Salinas E, Youssoufian H, Moore KN, Lustgarten S, O'Malley DM, Van Gorp T, Grisham RN. Efficacy and Safety of Avutometinib +/- Defactinib in Recurrent Low-Grade Serous Ovarian Cancer: Primary Analysis of ENGOT-OV60/GOG-3052/RAMP 201. J Clin Oncol. 2025 Sep;43(25):2782-2792. doi: 10.1200/JCO-25-00112. Epub 2025 Jul 11. PMID 40644648
- [Derived] Grisham R, Monk BJ, Van Nieuwenhuysen E, Moore KN, Fabbro M, O'Malley DM, Oaknin A, Thaker P, Oza AM, Colombo N, Gershenson D, Aghajanian CA, Choi CH, Lee YC, Mirza MR, Coleman RL, Cobb L, Harter P, Lustgarten S, Youssoufian H, Banerjee S. GOG-3097/ENGOT-ov81/GTG-UK/RAMP 301: a phase 3, randomized trial evaluating avutometinib plus defactinib compared with investigator's choice of treatment in patients with recurrent low grade serous ovarian cancer. Int J Gynecol Cancer. 2025 Nov;35(11):101832. doi: 10.1136/ijgc-2024-005919. Epub 2025 Apr 19. PMID 39375168